CLINICAL TRIAL: NCT02512029
Title: 18F-AV-1451 PET Imaging in Subjects With Subacute Traumatic Brain Injury
Brief Title: 18F-AV-1451 PET Imaging in TBI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A12
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBI Subjects (Experimental): Subjects with history of recent subacute Traumatic Brain Injury (TBI) will receive a single IV injection, 370 megabecquerel (MBq) [10 millicurie (mCi)] of 18F-AV-1451 2 to 6 weeks following injury. They will return for a follow-up injection approximately 6 months following injury.
  Interventions: Drug: 18F-AV-1451
- Control (Experimental): Cognitively healthy volunteer subjects will receive a single IV injection, 370 megabecquerel (MBq) [10 millicurie (mCi)] of 18F-AV-1451.
  Interventions: Drug: 18F-AV-1451

INTERVENTIONS:
Drug: 18F-AV-1451
  Other Names: [F-18]T807

SUMMARY:
This study will evaluate imaging characteristics of 18F-AV-1451 in subjects with subacute traumatic brain injury.

ELIGIBILITY:
TBI Subjects

Inclusion Criteria:

TBI Subjects

* Subjects that have consented and are currently enrolled in either Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI), Evaluation, Pathogenesis, and Outcome of Subjects with or Suspected Traumatic Brain Injury Protocol Number: CNS: 10-N-N122, or Evaluation and Diagnosis of Potential Research Subjects with Traumatic Brain Injury (TBI): Protocol Number: 11-N-0084
* History of having sustained a TBI < 6 weeks prior to enrollment
* Can tolerate PET and MRI scan procedures

Control Subjects

* MMSE ≥ 28
* No significant history of cognitive impairment
* No prior history of TBI
* Can tolerate PET and MRI scan procedures

Exclusion Criteria:

* Have behavior dysfunction that is likely to interfere with imaging
* Are claustrophobic or otherwise unable to tolerate the imaging procedure
* Have current clinically significant cardiovascular disease, or clinically significant abnormalities on screening ECG
* A history of additional risk factors for Torsades de Pointes (TdP) or are taking drugs that are known to cause QT-prolongation
* Have a current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception
* Have had a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to the 18F-AV-1451 imaging session
* Have current alcohol dependence or alcohol dependence within the past 1 year
* Are currently participating in another interventional clinical trial
* Have evidence of a penetrating brain injury
* Have participated in contact sports in college or after high school age

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
TBI Biomarker Analysis | 75-105 minutes postinjection
  18F-AV-1451 uptake will be compared in subjects with TBI and controls.
Relationship Between Clinical Presentation and Tau Deposition (MMSE) | 75-105 minutes postinjection
  The relationship between 18F-AV-1451 uptake and clinical measures using Mini-Mental State Examination (MMSE).
Change in tau deposition over time | 6 months
  Assess the rate of change of tau deposition as measured by 18F-AV-1451 uptake over time.
Relationship Between Clinical Presentation and Tau Deposition (BIS-11) | 75-105 minutes postinjection
  The relationship between 18F-AV-1451 uptake and clinical measures using Barratt Impulsivity Scale 11 (BIS-11)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (1):
- NIH Clinical Center, Bethesda, Maryland, United States